CLINICAL TRIAL: NCT05997654
Title: Evaluation of the Safety and Effectiveness of the Investigational Product in Improvement of the Appearance of Wrinkles and General Aspect of the Skin - Clinical, Instrumental and Subjective Study
Brief Title: Evaluation of the Safety and Effectiveness of the Investigational Product in Improvement of the Appearance of Wrinkles and General Aspect of the Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Silimed Industria de Implantes Ltda (Industry)
Collaborators: Medcin Instituto da Pele Ltda (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EN22-0300-01
Record Dates: First submitted 2023-07-21; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Skin Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Instrumental procedures and safety and efficacy assessments (Experimental): Group I: 23 participants who will undergo instrumental procedures, perceived efficacy questionnaires and clinical assessments of safety and efficacy.
  Group II: 10 participants who will only perform perceived efficacy questionnaires and clinical assessments of safety and efficacy.
  Interventions: Device: MEDGEL ANTIAGE

INTERVENTIONS:
Device: MEDGEL ANTIAGE — The MEDGEL ANTIAGE is a medical grade silicone plate, biocompatible.

SUMMARY:
The study investigates the safety and effectiveness of SILIMED® brand MEDGEL ANTIAGE with indication for improvement of the appearance of wrinkles and general aspects of the skin.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged between 30 and 55 years old;
* Participants with all skin types (normal, dry, combination and oily);
* Participants with mild to moderate signs of aging, according to Lanier's classification;
* Participants with melanic and/or vascular dark circles;
* Participants with bags around their eyes;
* Users of products from the same category;
* Intact skin in the product analysis region (face);
* Participants who agree NOT to use any other topical products on the test area during the study period;
* Agreement to comply with the trial procedures and to attend the clinic on the specified days and times;
* Understand, consent and sign the informed consent.

Exclusion Criteria:

* Participants diagnosed with COVID-19 in the last 4 weeks or showing symptoms such as fever, dry cough, tiredness, body aches or other discomfort;
* Pregnancy/lactation or intention to become pregnant during the study period;
* Use of the following topical or systemic medications: immunosuppressants, antihistamines, non-steroidal anti-inflammatory drugs, and corticoids up to 30 days before selection or considering immunosuppressants, the interval should be 3 months before selection;
* Atopic or allergic history of health products;
* Pathologies and/or active skin lesions (local and/or disseminated) in the assessment area;
* Skin marks in the experimental area that interfere with the evaluation of possible skin reactions (vascular malformations, scars, increased hairiness, large amounts of nevus, sunburn);
* Immunosuppression by drugs or active diseases;
* Decompensated endocrinopathies;
* Participants with known congenital or acquired immunodeficiency;
* Relevant medical history or current evidence of alcohol or other drug abuse;
* Known history or suspected intolerance to products in the same category
* Intense sun exposure up to 15 days before the assessment;
* Aesthetic or dermatological treatment in the evaluation area up to 04 weeks before selection;
* Professionals directly involved in carrying out this study;
* Other conditions considered by the evaluating physician as reasonable for disqualification from participating in the study. If yes, it should be described in observation in the clinical record

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2023-05-17 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2023-07-06 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events | 28 days
  Absence of risk of irritation and capture sensations of discomfort in the studied population through dermatological clinical evaluations before and after continuous use of the experimental product.

SECONDARY OUTCOMES:
Change in skin hydration | 1h, 2h, 4h, 6h, 8h and after 28 days
  Evaluate the effectiveness in changing skin hydration, through measurements by the CORNEOMETER® equipment after 1h, 2h, 4h, 6h and 8h of product contact with the skin and after 28 days of continuous use.
% of change in melanic and vascular dark circles | Before use and after 28 days of continuous use
  Evaluate the effectiveness of the investigational product in changing % of melanic and vascular dark circles through photographic recording by the VISIA® equipment and image analysis by Image Pro Plus, before use (D0) and after continuous use (D28).
Change in skin firmness and elasticity | Before use and after 28 days of continuous use
  Evaluate the effectiveness of the investigational product in changing skin firmness and elasticity through instrumental measurements by the CUTOMETER® equipment, before use (D0) and after continuous use (D28).
Change in furrows and wrinkles depth | Before use and after 28 days of continuous use
  Evaluate the effectiveness of the investigational product in changing furrows and wrinkles depth through photographic records by the PRIMOS® equipment, before use (D0) and after continuous use (D28).
Satisfaction assessed by a subjective questionnaire using a standardized 05-point scale | Before use and after 28 days of continuous use
  Evaluate the satisfaction with the investigational product from the point of view of the target population through a subjective questionnaire using a standardized 05-point scale answered before (D0) and after continuous use (D28).

CONTACTS AND LOCATIONS:
Locations (1):
- Medcin Instituto da Pele Ltda, Osasco, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No